CLINICAL TRIAL: NCT04611711
Title: An Evaluation of the Effectiveness and Safety of Decitabine Combined With TQB2450 Injection (PD-L1 Monoclonal Antibody) or Decitabine + Anlotinib Combined With TQB2450 Injection in the Treatment of PD-1 Monoclonal Antibody-resistant Digestive System Tumors I /Phase II Clinical Study
Brief Title: Phase I/II Clinical Study of Decitabine Combined With TQB2450 Injection or Decitabine + Anlotinib Combined With TQB2450 Injection in the Treatment of PD-1 Monoclonal Antibody-resistant Digestive System Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-I/II-01
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-09

CONDITIONS: Patients With Digestive System Tumors Resistant to PD-1 Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- decitabine＋ TQB2450 injection (PD-L1 monoclonal antibody) (Other): Decitabine (10mg ivgttqd, d1-5) combined with TQB2450 injection (1200mg ivgtt, d5)
  Interventions: Drug: decitabine＋ TQB2450 injection
- decitabine + anlotinib ＋ TQB2450 injection (PD-L1 monoclonal antibody) (Other): Decitabine and Anlotinib (decitabine 10mg ivgtt qd, d1-5; Anlotinib 8mg po.qd, d5-18) combined with TQB2450 injection (1200mg ivgtt, d5), using the traditional 3+3 experimental design (First enroll 3 subjects. If 1 case of DLT is observed, 3 more subjects need to be added to the same dose group to further evaluate the toxicity) to observe DLT to evaluate MTD. The trial starts from the 8mg dose of Anlotinib Start.
  Interventions: Drug: decitabine＋ TQB2450 injection＋Anlotinib

INTERVENTIONS:
Drug: decitabine＋ TQB2450 injection — "Real low-dose epigenetics drugs (decitabine) can reverse the resistance of PD-1 inhibitors by re-regulating the immune microenvironment.
  TQB2450 is a humanized monoclonal antibody targeting PD-L1, which prevents PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, so as to restore the activity of T cells and thereby enhance the immune response, and has the potential to treat various types of tumors."
  Arms: decitabine＋ TQB2450 injection (PD-L1 monoclonal antibody)
Drug: decitabine＋ TQB2450 injection＋Anlotinib — "Real low-dose epigenetics drugs (decitabine) can reverse the resistance of PD-1 inhibitors by re-regulating the immune microenvironment.
  TQB2450 is a humanized monoclonal antibody targeting PD-L1, which prevents PD-L1 from binding to the PD-1 and B7.1 receptors on the surface of T cells, so as to restore the activity of T cells and thereby enhance the immune response, and has the potential to treat various types of tumors.
  Anlotinib Hydrochloride is a multi-target receptor tyrosine kinase inhibitor with significant inhibitory activity against angiogenesis related kinases (VEGFR1/2/3, FGFR1/2/3, etc.) and other tumor cell proliferation-related kinases (PDGFR /, C-Kit, RET, etc.), which can play a dual role in anti-tumor angiogenesis and tumor growth inhibition. "
  Arms: decitabine + anlotinib ＋ TQB2450 injection (PD-L1 monoclonal antibody)

SUMMARY:
This clinical study focused on patients with digestive system tumors resistant to PD-1 inhibitors, and explored the reversal resistance of epigenetic drugs (decitabine) and TKI drugs (anlotinib) in this part of patients.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written informed consent;
* Age: 18-70 years old;
* No gender limitation;
* Digestive system malignant tumor diagnosed by pathology;
* Previously received PD-1 monoclonal antibody Or the combination therapy fails;
* There is at least one measurable lesion (according to the RECIST1.1 standard) or an unmeasurable lesion that can be evaluated, and the imaging diagnosis is ≤21 days from the selection time；
* The expected survival period is ≥3 months;
* General physical status (ECOG) 0-1;
* Sufficient bone marrow hematopoietic function (within 7 days); normal liver and kidney function (within 14 days)；
* Heart, lung, kidney, and liver functions are generally normal.

Exclusion Criteria:

* People who are currently receiving other effective treatments;
* Patients who have been treated with anti-vascular TKI drugs in the past;
* Patients who have participated in other clinical trials within 4 weeks before enrollment;
* Allergic to study drugs;
* Those without measurable tumor lesions, such as body cavity effusion or diffuse infiltration of organs;
* Those with measurable lesions that have received radiotherapy.
* Patients with other primary malignant tumors other than digestive system tumors at the same time, except for early solid tumors that have been cured for more than 1 year;
* Clinically significant cardiovascular diseases, such as heart failure (NYHAIII-IV), are not controlled A history of coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or myocardial infarction within the past 1 year;
* Neurological or mental disorders that affect cognitive ability, including central nervous system metastasis;
* Existed within 14 days before enrollment Active severe clinical infections (>grade 2 NCI-CTCAE version 5.0), including active tuberculosis;
* Known or self-reported HIV infection or active hepatitis B or C;
* Uncontrolled Systemic diseases, such as poorly controlled diabetes;
* A history of interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease on baseline chest X-ray/CT;
* Keratitis , Ulcerative keratitis or severe dry eye;
* Known hypersensitivity or allergic reaction to any component of the study drug;
* Pregnancy (determined by serum β-chorionic gonadotropin test) or breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Objective response rate refers to the percentage of complete (CR) or partial response (PR) subjects determined by the investigator based on RECIST 1.1 or iRECIST (CR under iRECIST criteria, PR can occur after imaging disease progression).

SECONDARY OUTCOMES:
Overall survival (OS) | up to 48 weeks
  Overall survival defined as the time from enrollment to death from any cause.